CLINICAL TRIAL: NCT03469583
Title: Study of the Drug Interaction of EYP001a With Entecavir in Healthy Subjects
Brief Title: Drug Drug Interaction Study for EYP001 With Entecavir
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Enyo Pharma (Industry)
Collaborators: CPR Pharma Services Pty Ltd, Australia (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: EYP001-104
Record Dates: First submitted 2018-01-29; First posted 2018-03-19 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — entecavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- EYP001 dose1 (Experimental): EYP001 capsules by mouth
  Interventions: Drug: EYP001
- Entecavir 1mg (Active Comparator): 2 tablets of 0.5mg, by mouth
  Interventions: Drug: Entecavir 1 MG
- EYP001 dose 1 + Entecavir 1mg (Experimental): EYP001 capsules and 2 tablets of Entecavir 0.5mg by mouth
  Interventions: Drug: EYP001; Drug: Entecavir 1 MG

INTERVENTIONS:
Drug: EYP001 — EYP001 self administered capsules, morning, with non carbonated water
  Other Names: EYP001a
  Arms: EYP001 dose 1 + Entecavir 1mg; EYP001 dose1
Drug: Entecavir 1 MG — Entecavir self administered tablets, morning, with non carbonated water
  Other Names: ETV
  Arms: EYP001 dose 1 + Entecavir 1mg; Entecavir 1mg

SUMMARY:
This is a Phase 1, single-center, open-label, three subsequent dosing periods study to evaluate the drug-drug-interaction (DDI), pharmaco-kinetics (PK) and pharmacodynamics (PD), safety, and tolerability of a single dose of EYP100a combined with ETV in healthy men and women dosed in the morning under fasted conditions.

DETAILED DESCRIPTION:
This is a Phase 1, single-center, open-label, three consecutive dosing periods study to evaluate the drug-drug interaction, PK, safety, tolerability and PD of a single dose of EYP100a combined with ETV in healthy men and women. Sixteen (16) adult male and female healthy participants 18 to 60 years of age inclusive are planned to participate in the study. Women of childbearing potential will be eligible to participate if she is non pregnant or non lactating and willing to use adequate contraception.

All participants in the study will be monitored for safety after administration of the last dose of investigational product and with a follow up visit. The DDI, PK, PD, safety and tolerability of EYP001a and ETV will be assessed based on plasma-concentration profiles of EYP001a and ETV, FXR related PD markers and the types and frequency of treatment-emergent adverse events (TEAEs) reported, concomitant medication usage, and changes from baseline in physical examination (PE), vital signs, electrocardiogram (ECG), and standard clinical laboratory tests.

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided written consent
* In the investigator's opinion, the subject is able to understand and comply with protocol requirements, instructions, and study restrictions and is likely to complete the study as planned
* Subject is in good health as deemed by the investigator, based on the findings following a medical evaluation, including medical history, physical examination, laboratory tests and single ECG
* Male or female, 18-60 years of age inclusive
* Body mass index 18.0-35.0 kg/m2, inclusive. The minimum weight is 50 kg, the maximum is 115 kg.
* A female subject is eligible to participate in this study if:

  1. She is of non-childbearing potential (defined as females with a documented tubal ligation, bilateral oophorectomy or hysterectomy) or postmenopausal (defined as 12 months of spontaneous amenorrhea and follicle stimulating hormone level within the laboratory's reference range for postmenopausal females). A post-menopausal female receiving hormone replacement therapy (HRT) other than hormone replacement patches who is willing to discontinue hormone therapy 28 days before study drug dosing and agrees to remain off hormone replacement therapy for the duration of the study may be eligible for study participation. A post menopausal female using Hormone Replacement patches who is willing to discontinue the patch 48 hours before Check in on Day -1 and until the completion of her End of Study visit is eligible for study participation
  2. She is of childbearing potential and is non pregnant or non lactating and willing to use adequate contraception from screening until 6 months after the End of Study visit. Adequate contraception is defined as a progesterone only intra uterine device combined with at least 1 of the following forms of contraception: a diaphragm or cervical cap, or a condom. Also, total abstinence in accordance with the lifestyle of the participant. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception
  3. She is of childbearing potential and is non pregnant or non lactating and taking the combined oral contraceptive pill and willing to discontinue the combined oral contraceptive pill 7 days prior to check in on Day -1 and until the completion of her End of Study visit and use adequate contraception from the day of cessation. Adequate contraception is defined as a diaphragm or cervical cap together with a condom. Also, total abstinence in accordance with the lifestyle of the participant is acceptable. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.
* If male, subject is surgically sterile or practicing required forms of birth control until 6 months after the last dose of the study drug(s). Males must agree to refrain from sperm donation from check-in through 6 months after the last dose of the study drug(s)
* Subject does not use nicotine or nicotine-containing products during study participation.

Exclusion Criteria:

* Subject is mentally or legally incapacitated, has significant emotional problems at the time of prestudy (screening) visit or expected during the conduct of the study or has a history of a clinically significant psychiatric disorder over the last 5 years.
* Subject has a history of any illness that, in the opinion of the investigator, would confound the objectives or results of the study or poses an additional risk to the subject by their participation in the study
* Subject has an estimated creatinine clearance of ≤ 80 mL/min based on the Cockcroft-Gault equation; subjects who have an actual or estimated creatinine clearance within 10% of 80 mL/min may be enrolled in the study at the discretion of the investigator.
* Pregnant or nursing (lactating) females, confirmed by a positive human chorionic gonadotropin laboratory test or females contemplating pregnancy. Men whose female partners are pregnant or contemplating pregnancy from the date of screening until 6 months after their last dose of study drugs
* Clinically significant cardiovascular, respiratory, skeletal, renal, gastrointestinal, hematologic, hepatic, immunological, neurologic, endocrine, genitourinary abnormalities or disease or any other medical illness as determined by the investigator or Sponsor's Medical Monitor
* Subject has a history of malignancy except completely excised basal cell carcinoma or squamous cell carcinoma of the skin
* Subject lacks or has poor peripheral venous access
* Positive screening result for hepatitis B, hepatitis C and/or HIV serology
* Any condition that, in the opinion of the investigator, would compromise the study's objectives or the well-being of the subject or prevent the subject from meeting the study requirements
* Clinically significant abnormal ECG findings. Particularly, a history or family history of prolonged QT syndrome (eg, torsades de pointes) or sudden cardiac death.
* ECG with PR >220 ms, QRS >120 ms, QTcF >450 ms, as assessed by 12-lead ECG at the screening visit
* Subject has had major surgery, or clinically significant blood loss or elective blood donation of significant volume (ie, >500 mL) within 60 days of first dose of study drug; >1 unit of plasma within 7 days of first dose of study drug
* Abnormal heart rate, respiratory rate, temperature or blood pressure values outside of the normal range (evaluated in a semi-recumbent or recumbent position after 5 minutes of rest). One repeat measurement after an additional 5 minutes of rest is permitted
* Evidence of active infection
* Unwilling to abstain from alcohol for at least 48 hours prior Day 1 through to the end of the study
* History of regular alcohol intake >7 units per week of alcohol for females and >14 units per week for males (one unit is defined as 10 g alcohol) within 3 months of the screening visit
* The subject has a positive screening for drugs of abuse on Day -1 or Day 9 at check in prior to the start of the confinement periods.
* The use of concomitant medications, including prescription, over the counter medications, and herbal medications (such as St. John's Wort [Hypericum perforatum]) (except for HRT patches, combined oral contraceptive pills and Progesterone IUD) within 30 days prior to the first dose of study medication is excluded, unless approved by the Sponsor's Medical Monitor. Occasional use of ibuprofen/paracetamol (acetaminophen) is permitted
* Subject has received an investigational drug (including investigational vaccines) or used an invasive investigational medical device within 90 days before the planned study drug
* Subject has a history of significant* multiple and/or severe allergies
* Hypersensitivity to the active substances or to any of the excipients of EYP001a and or ETV
* Abnormal biochemistry or hematology laboratory results obtained at screening determined to be clinically significant by the Investigator. Screening ALT, AST, GGT, albumin, and total bilirubin must be within normal ranges. Creatine kinase >1.5 x ULN is exclusionary
* Unwillingness or inability to comply with the study protocol for any other reason.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — 8 males and 8 females.
Enrollment: 16 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2018-06-20 (Actual); Study Completion 2018-07-20 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve | 24 hrs
  Area under the concentration-time curve from time 0 to 24 hours

SECONDARY OUTCOMES:
Adverse events | Day 1 to Day 12
  Treatment emergent adverse events
Concentration maximum (peak) | Day 1, Day 3 and Day 10
  highest concentration of EYP001 and ETV after dosing
Volume of distribution (Vz/F) | 8 days
  Pharmacokinetic endpoints
Time to maximum concentration (Tmax) | 8 days
  Pharmacokinetic endpoints
Terminal Elimination Rate Constant (kel) | 8 days
  Pharmacokinetic endpoints
Terminal half-life (t1/2) | 8 days
  Pharmacokinetic endpoints
Terminal clearance (CL/F) | 8 days
  Pharmacokinetic endpoints
C4 and FGF19 | Day 1, Day 3 and Day 10
  C4 (7αhydroxy-4-cholesten-3- one) and fibroblast growth factor 19 (FGF19) are PD Marker of FXR engagement

CONTACTS AND LOCATIONS:
Overall Officials: Angela Molga, M.D. FRACP, Principal Investigator — CMAX - Clinical Research Pty Ltd, Level 5, 18a North Terrace, Adelaide, South Australia, 5000, Australia
Locations (1):
- Cmax Clinical Research Pty Ltd, Adelaide, South Australia, Australia